CLINICAL TRIAL: NCT07117084
Title: Imaging Markers of High-Risk Plaque Phenotype for Predicting Post-PCI Outcomes (IMPACT-PCI) Study: A Multicenter Cohort Study Based on Coronary CT Angiography
Brief Title: Imaging Markers of High-Risk Plaque Phenotype for Predicting Post-PCI Outcomes
Acronym: IMPACT-PCI
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Bin Lu, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: IMPACT-PCI study; 2024-2586 (Other: Fuwai Hospital)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention (PCI); Atherosclerosis of Coronary Artery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCTA-PCI Cohort: Patients who underwent coronary CT angiography followed by PCI within 30 days.
  Interventions: Diagnostic Test: CCTA-derived Plaque Quantification

INTERVENTIONS:
Diagnostic Test: CCTA-derived Plaque Quantification — Quantitative analysis of coronary plaque features based on coronary CT angiography using semi-automated software.

SUMMARY:
Despite the widespread use of stents, previous studies have shown that stent implantation mainly relieves symptoms but may not significantly improve long-term outcomes in patients with stable coronary artery disease. Identifying the types of plaques that are most likely to benefit from stenting is essential for improving personalized treatment. This study explores whether coronary computed tomography angiography (CCTA)-derived imaging biomarkers of coronary plaques are associated with increased risk of adverse outcomes after percutaneous coronary intervention (PCI). Around 2,000 patients who underwent CCTA followed by stent placement were included. Advanced software was used to quantify plaque inflammation and composition. Findings from this research may help guide personalized treatment strategies in patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18 years or older;
2. patients who underwent clinically indicated PCI within 30 days following CCTA;
3. CCTA demonstrating the presence of coronary atherosclerotic plaque.

Exclusion Criteria:

1. patients whose PCI within 30 days after CCTA was performed on an emergency basis;
2. elevated cardiac troponin levels within the 3 months preceding PCI;
3. inadequate CCTA image quality;
4. balloon-only or mixed stent/balloon PCI strategies;
5. PCI for non-atherosclerotic lesions (e.g., in-stent restenosis, spontaneous coronary dissection);
6. history of coronary artery bypass grafting;
7. heart failure;
8. non-ischemic cardiomyopathy;
9. significant valvular heart disease;
10. refractory hypertension;
11. persistent atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent clinically indicated PCI within 30 days after coronary CT angiography.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | From the date of PCI until December 2024 (minimum 2-year follow-up)
  Composite of cardiovascular death, non-fatal myocardial infarction, repeat revascularization, and hospitalization for unstable angina.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lu, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (3):
- China (3):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Tai'an Central Hospital, Tai’an, Shandong
  - Weifang People's Hospital, Weifang, Shandong

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional data privacy policies and lack of data-sharing agreements.